CLINICAL TRIAL: NCT07267923
Title: Investigation of the Acute Effects of Traditional and Functional Inspiratory Muscle Training on Muscle Oxygenation in Chronic Obstructive Pulmonary Disease
Brief Title: Investigation of the Acute Effects of Traditional and Functional IMT on Muscle Oxygenation in COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/489
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; inspiratory muscle training; functional inspiratory muscle training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This study uses a crossover design with a single participant group, in which all participants receive both exercise interventions. Each participant will undergo one baseline assessment prior to any intervention. On separate days, participants will complete two different inspiratory muscle training (IMT) interventions: conventional IMT and functional IMT. A standardized outcome assessment is performed immediately after each intervention session, resulting in a total of three measurement time points (pre-intervention, post-conventional IMT, and post-functional IMT). Outcomes obtained at these three time points will be compared to determine the acute effects and relative impact of each training modality.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic Obstructive Pulmonary Disease (Experimental)
  Interventions: Other: Traditional inspiratory muscle training; Other: Functional inspiratory muscle training (IMT)

INTERVENTIONS:
Other: Traditional inspiratory muscle training — Traditional inspiratory muscle training is a form of training performed using a resistive breathing device that provides resistance to the muscles involved in inspiration. Inspiratory muscle training will be performed using a portable pressure-threshold device (POWERbreathe Classic IMT - Light Resistance). IMT will be administered in a seated position with upper extremities supported and the upper chest/shoulders relaxed. The training procedure will be explained to each participant and performed for 15 minutes at 40% of the maximal inspiratory pressure (MIP).
Other: Functional inspiratory muscle training (IMT) — Functional inspiratory muscle training (IMT) is defined as inspiratory muscle training performed while maintaining core stabilization and postural control. Functional IMT consists of a warm-up period, core exercises, dynamic trunk activation combined with upper extremity movements, postural control exercises, and a cool-down period. The participant performs these exercises simultaneously with inspiratory muscle training.

SUMMARY:
This study aims to compare the effects of functional and conventional inspiratory muscle training (IMT) on post-exercise muscle deoxygenation in individuals with Chronic Obstructive Pulmonary Disease (COPD). Participants will complete both training modalities on separate days. A 2-minute walk test (2MWT) will be performed baseline, and after each session. Muscle oxygenation (SmO₂) will be assessed using near-infrared spectroscopy . Dyspnea and fatigue will be evaluated with the Modified Borg Scale, and heart rate and oxygen saturation (SpO₂) will be measured by pulse oximetry. Measurements will be recorded before, after training and at the end of the walking test.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Having a diagnosis of COPD,
* Being in stage II-III according to the GOLD classification,
* Being able to mobilize independently.

Exclusion Criteria:

* Having a recent exacerbation or complication requiring hospitalization,
* Having had a respiratory tract infection within the past month,
* Having any disease or medical condition that prevents participation in exercise, -Having cognitive impairment (a score of <24 on the Mini-Mental Test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Muscle oxygenation levels (SmO₂) | 1. day - baseline measurement-before and after 2MWT , 1. day- before and after IMT and after 2MWT 2. day- before and after FIMT and after 2MWT
  Muscle oxygenation (SmO₂) will be assessed using near-infrared spectroscopy .

SECONDARY OUTCOMES:
Fatigue | 1. day - baseline measurement-before and after 2MWT , 1. day- before and after IMT and after 2MWT 2. day- before and after FIMT and after 2MWT
  Fatigue will be assessed before and after the walking test using the Borg scale. The scale is scored from 0 to 10, with 0 being no fatigue and 10 being extreme fatigue.
Dyspnea | 1. day - baseline measurement-before and after 2MWT , 1. day- before and after IMT and after 2MWT 2. day- before and after FIMT and after 2MWT
  Dyspnea severity will be assessed using the Modified Borg Scale. It consists of ten items that describe the severity of dyspnea according to degree. The scale is scored from 0 (no shortness of breath) to 10 (very severe).
Heart rate | 1. day - baseline measurement-before and after 2MWT , 1. day- before and after IMT and after 2MWT 2. day- before and after FIMT and after 2MWT
  Heart rate value will be measured with a pulse oximeter.
Saturation (SPO2) | 1. day - baseline measurement-before and after 2MWT , 1. day- before and after IMT and after 2MWT 2. day- before and after FIMT and after 2MWT
  Saturation values will be measured with a pulse oximeter.
hemoglobin | 1. day - baseline measurement-before and after 2MWT , 1. day- before and after IMT and after 2MWT 2. day- before and after FIMT and after 2MWT
  The hemoglobin value of muscle tissue will be measured using the near infrared spectroscopy (NIRS) method.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Faculty of Physiotherapy and Rehabilitation, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No